CLINICAL TRIAL: NCT07108023
Title: A Prospective Study of the Spectrum of Haematological Disorders in Patients With Extrahepatic Portal Vein Obstruction
Brief Title: Hematological Disorders in EHPVO Patients
Acronym: EHPVO-HEM
Status: Not yet recruiting | Type: Observational
Sponsor: Rahab Nady (Other)
Responsible Party: Sponsor-Investigator, Rahab Nady, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: EHPVO-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Extrahepatic Portal Vein Obstruction (EHPVO); Thrombophilia; Myeloproliferative Neoplasms (MPN); Antiphospholipid Syndrome (APS); Paroxysmal Nocturnal Hemoglobinuria (PNH); Thrombocytopenia; Anemia; Leukopenia
Keywords: Portal vein thrombosis; EHPVO; Hypersplenism; Hematological disorders; Coagulation profile; Liver function tests; CBC; JAK2 mutation; Thrombosis in MPN; Cross-sectional study
MeSH Terms: conditions — Thrombophilia; Myeloproliferative Disorders; Antiphospholipid Syndrome; Hemoglobinuria, Paroxysmal; Thrombocytopenia; Anemia; Leukopenia; Hypersplenism; Hematologic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EHPVO Patients: Patients diagnosed with extrahepatic portal vein obstruction (EHPVO) based on imaging (Doppler ultrasound, CT, or MRI) and with preserved liver function. This group will be assessed for hematological abnormalities, including cytopenias and coagulation disturbances, using retrospective laboratory data.
  Interventions: Other: No intervention (Observational Study)

INTERVENTIONS:
Other: No intervention (Observational Study) — This is a retrospective observational study with no assigned intervention. Data will be collected from patient medical records only

SUMMARY:
This study focuses on patients who have a condition called extrahepatic portal vein obstruction (EHPVO), where a blood clot blocks the portal vein outside the liver. This blockage can cause problems like an enlarged spleen, bleeding from swollen veins in the digestive system, and low blood cell counts. Many of these patients may have hidden blood disorders that increase the risk of clotting, such as myeloproliferative neoplasms (MPNs), antiphospholipid syndrome (APS), or paroxysmal nocturnal hemoglobinuria (PNH). This study will collect and analyze blood test results-such as complete blood count (CBC), liver function tests (LFTs), and clotting tests-from patients with EHPVO. The aim is to find patterns that may suggest an underlying blood disorder, even if the patient doesn't show obvious symptoms.By understanding these patterns early, doctors may be able to diagnose and treat the root causes of clotting in these patients more accurately, helping prevent complications and improve outcomes.

DETAILED DESCRIPTION:
Extrahepatic portal vein obstruction (EHPVO) is a non-cirrhotic cause of portal hypertension that results from a thrombotic blockade in the portal vein outside the liver. The preserved hepatic parenchyma distinguishes EHPVO from intrahepatic causes of portal hypertension. However, complications like variceal bleeding, hypersplenism, and splenomegaly remain common. Hematological abnormalities frequently observed in EHPVO include thrombocytopenia, anemia, and leukopenia, often attributed to hypersplenism. Yet, in a subset of patients, especially those with concurrent myeloproliferative neoplasms (MPNs), these cytopenias may be masked due to increased production of blood elements. Coagulation profiles may also show subtle abnormalities or evidence of underlying thrombophilia.A growing body of literature suggests a strong association between EHPVO and underlying prothrombotic conditions such as MPNs (often linked to JAK2V617F mutation), antiphospholipid syndrome (APS), and paroxysmal nocturnal hemoglobinuria (PNH).

Early identification of these disorders may significantly impact clinical management, prognosis, and long-term surveillance. The current study is a cross-sectional observational analysis aiming to investigate the hematological spectrum in patients with EHPVO at Assiut University Hospital. Data will be collected retrospectively from medical records, including CBC with differential, liver function tests, coagulation parameters, and specific thrombophilia workups when available. The primary objective is to correlate these laboratory findings with underlying hematological disorders. Secondary aims include evaluating the association between these abnormalities and clinical outcomes such as variceal bleeding, transfusion needs, and prognosis. The study may offer valuable insights into risk stratification and highlight the importance of thrombophilia screening in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older . Diagnosis of extra hepatic portal vein obstruction based on imaging ( Doppler, CT , MRI ) preserved liver function . Available complete medical records including CBC , LFTs and coagulation profile .

Exclusion Criteria:

* Patients with cirrhosis or intrahepatic portal hypertension • Incomplete or missing medical records • Patients with known hematologic malignancies or undergoing chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with EHPVO between 2020 and 2024 in a tertiary care hospital in Cairo. Data will be collected retrospectively from medical records
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of hematological disorders in EHPVO patients | Over a retrospective period from 2020 to 2024
  The proportion of EHPVO Patients showing hematological disorders including cytopenias ( thrombocytopenia , anemia , leukopenia ) and coagulation disturbances based on retrospective laboratory data
Frequency of hematological disorders in EHPVO patients | Over a retrospective period from 2020 to 2024

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Q Professor of internal medicine, Principal Investigator — Assiut University; Maha M Dr Maha Mohamed Abdelaziz, Dr at Internal medicine, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including complete blood count (CBC), liver function tests (LFTs), and coagulation profile results, will be shared. No personally identifiable information will be included.
Supporting Information: Study Protocol
Time Frame: IPD and supporting documents will be available starting 6 months after publication of the primary results and will remain available for up to 5 years after publication.
Access Criteria: Access to the de-identified individual participant data (IPD), including CBC, LFTs, and coagulation profiles, will be granted to qualified researchers for academic and non-commercial purposes.
  Requests should be submitted to the Principal Investigator and will be reviewed on a case-by-case basis. A data use agreement may be required before access is granted.

REFERENCES:
- See also: Related Info — https://emedicine.medscape.com/article/182425-overview?form=fpf